CLINICAL TRIAL: NCT06424275
Title: Prostate Cancer Awareness and Initiative for Screening in the European Union
Acronym: PRAISE-U
Status: Enrolling by invitation | Type: Observational
Sponsor: European Association of Urology Research Foundation (Other)
Collaborators: Erasmus Medical Center (Other); European Randomised Study of Screening for Prostate Cancer (Unknown); Region MidtJylland Denmark (Other); Institute of Health Information and Statistics of the Czech Republic (Other Government); UMC Utrecht (Other); EUROPEAN CANCER ORGANISATION (Unknown); Dolnośląskie Centrum Onkologii, Pulmonologii i Hematologii (Unknown); Narodowy Instytut Zdrowia Publicznego (Unknown); Conselleria de Sanidade de Galicia (Unknown); Althaia Xarxa Assistencial Universitària de Manresa (Other); Vastra Gotaland Region (Other Government); Region Skane (Other); National Cancer Institute (NCI) (NIH); University Ghent (Other); Health Service Executive, Ireland (Other); Estonian Urological Association (Unknown); University College Dublin (Other); WONCA Europe (Unknown); Movember Foundation (Other); International Agency for Research on Cancer (Other); European Society of Urogenital Radiology (Other); Europa UOMO (Unknown); Czech Urological Society (Unknown)
Responsible Party: Sponsor
Other Study IDs: 101101217
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; early detection of prostate cancer; cancer screening; risk-based algorithm
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Manresa, Spain: The pilot is run by the Althaia Foundation, driven by the director of primary care.
  Interventions: Diagnostic Test: Risk-based screening algorithm
- Region Galicia, Spain: The pilot is run by the Galician Healthcare Service (SERGAS), publicly funded healthcare system of Galicia, Spain.
  Interventions: Diagnostic Test: Risk-based screening algorithm
- Ireland: The pilot is run by the Health Service Executive, with University College Dublin as the academic institutional partner, in full support of the National Cancer Control programme (NCCP) and the National Screening Service (NSS) in Ireland
  Interventions: Diagnostic Test: Risk-based screening algorithm
- Poland: The pilot is run by the Lower Silesian Oncology, Pulmonology and Haematology Center. Subdivision of Urology with support from the National Institute of Public Health.
  Interventions: Diagnostic Test: Risk-based screening algorithm
- Lithuania: The pilot is run by the National Cancer Institute, where residents of the capital Vilnius region are served.
  Interventions: Diagnostic Test: Risk-based screening algorithm

INTERVENTIONS:
Diagnostic Test: Risk-based screening algorithm — Risk-based screening algorithm
  Other Names: PSA; Risk calculator; MRI; Biopsy

SUMMARY:
PRAISE-U was initiated on the 1st of April 2023 and is set to last for three years. This collaborative effort involves 25 institutions across 12 countries, all driven by a shared objective: to rationalize prostate cancer screening in Europe and enhance patient outcomes. PRAISE-U advocates for EU member states to offer exceptional clinical standards, incorporating cutting-edge personalized approaches to enable timely detection of prostate cancer in individuals who can benefit from early treatment. To assess the functionality, feasibility, and long-term viability of a risk-based algorithm, the consortium will collaborate with pilot sites in Spain, Poland, Ireland, and Lithuania.

DETAILED DESCRIPTION:
The project has several key deliverables that are instrumental in its success. In the early phase of the project, the consortium will prepare a living state-of-play document - a comprehensive review of diverse screening strategies for prostate cancer in the EU, as well their harm/benefit and cost effectiveness. At a later stage, clinical performance indicators of screening effectiveness will be established, and a protocol for implementation of population-based quality assured prostate cancer screening program will be developed. While the protocol will follow a standardized approach, it will also allow for flexibility to accommodate the unique characteristics of each country's healthcare system. The pilot studies will run for 12 months, and all collected data will be used to estimate pre-defined key performance indicators that will be included in the final report. This deliverable will be used to perform a thorough evaluation of how well the screening program worked during the pilot phase and how site characteristics and diagnostic algorithms are associated with performance. The reach, acceptability, and adoption of the screening programme, its cost-effectiveness, as well as attitudes of participants and physicians, will be the research outcomes of interest.

The project aims to have short-term and long-term effects on prostate cancer screening in EU member states. In the short-term (1-3 years), the focus is on advancing population-based risk-adapted prostate cancer screening and increasing awareness among key stakeholders. This will be achieved by providing evidence-based information on the benefits and drawbacks of risk-adapted screening, leading to improved knowledge and future endorsement by healthcare professionals. In the medium-term (4-9 years), the goal is to reduce costs by eliminating ineffective opportunistic screening and implementing an organized risk-based screening algorithm. Ultimately, in the long-term (10+ years), the project aims to decrease the burden of prostate cancer and improve quality of life by reducing mortality rates and the number of advanced/metastatic cases through effective screening practices. PRAISE-U is an important step in assessing how screening for prostate cancer may reduce the burden of the disease for every man in the European Union.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-69 years old.

Exclusion Criteria:

* Previous diagnosis of prostate cancer.
* Unable to provide written informed consent.
* Had prostate biopsy or MRI within the past six months.

Ages: 50 Years to 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy men aged 50-69 years old.
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of clinically significant prostate cancer in each pilot site (with clinically significant prostate cancer defined as ISUP grade group ≥2). | 1 year
Invitation coverage | 1 year
  The proportion of eligible individuals from the target population personally invited for screening within a given time frame.
Examination coverage | 1 year
  The proportion of eligible individuals from the target population who had the recommended screening test within a given time frame
Participation rate | 1 year
  The proportion of invited individuals who have undergone a screening test within a given time- frame following an active invitation.
Retention rate | 1 year
  The proportion of eligible individuals re-screened after a negative screening within a specified interval.
Test result | 1 year
  The results of the screening test.
PPV of screening test to detect any prostate cancer (6.1) and clinically significant prostate cancers (6.2) | 1 year
  The proportion of individuals who have histopathology confirmed PCa to all those who had positive test results (with PSA result of >3 ng/ml) (including healthy subjects who were incorrectly diagnosed to have prostate cancer)
PPV of screening test to detect any prostate cancer (6.1) and clinically significant prostate cancers (6.2) | 1 year
  The proportion of individuals who have histopathologically confirmed clinically significant PCa to all those who had positive test results (with PSA result of >3 ng/ml)
  (including healthy subjects who were incorrectly diagnosed as clinically significant PCa).
False positive rate to detect any PCa (7.1) and clinically significant PCa (7.2) | 1 year
  The proportion of screened individuals who received a positive screening result in which no cancer was detected after workup and diagnostic procedures.
False positive rate to detect any PCa (7.1) and clinically significant PCa (7.2) | 1 year
  The proportion of screened individuals who received a positive screening result in which no clinically significant cancer was detected after workup and diagnostic procedures.
Compliance with risk assessment | 1 year
  The proportion of individuals from the screened population undergoing risk assessment (as per protocol of the programme).
Compliance with further assessment | 1 year
  The proportion of individuals referred for diagnostic work up based on elevated PSA and risk assessment (as per protocol of the programme) attending all workup and diagnostic procedures assigned.
Detection rate of PCa | 1 year
  The proportion of individuals with a screen positive test who underwent further assessment with histopathologically proven cancer detected [expressed per 1,000 individuals screened].
Compliance with treatment | 1 year
  The proportion of individuals with cancer diagnosed within the screening program referred for treatment who initiated treatment (including active surveillance, when applicable).
Complications in screening procedure | 1 year
  The proportion of individuals reporting at least one complication incurred during the screening procedure.
Opportunistic testing | 1 year
  The proportion of individuals screened outside the population-based screening programme.
Cause-specific mortality | 1 year
  The mortality from prostate cancer (primary cause of death only) per 100,000 target population in a defined 12-month period
Crude Incidence rate | 1 year
  The number of new cases of PCa arising in a specified population (expressed per 100,000) within a time frame of 12-months.]
Interval cancer rate | 1 year
  The proportion of individuals with a negative screening test or a positive screening test but negative further assessment results who were diagnosed with prostate cancer prior to the next screening round.
Delay time | 1 year
  Time from PSA test sample collection to histopathological confirmation of a malignant diagnosis (further disaggregated by different procedures) to treatment initiation
Radiologist's assessment of MRI | 1 year
  Radiologist's assessment of MRI
Compliance with biopsy | 1 year
  Proportion of eligible men who underwent biopsy
Active surveillance | 1 year
  The proportion of patients recommended AS due to low/low-intermediate risk PCa who accepted and initiated AS.
Tumour grade distribution | 1 year
  Proportion of prostate cancers detected after positive screening test reported as ISUP grade (group) 1, 2, 3 and 4-5.

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik Van Poppel, Prof, Study Director — European Association of Urology and KULeuven; Monique J Roobol, Prof, Principal Investigator — Erasmus MC Cancer Institute Dep of Urology and European Association of Urology
Locations (5):
- University College Dublin, Dublin, Ireland
- National Cancer Institute, Vilnius, Lithuania
- Lower Silesian Oncology, Pulmonology and Hematology Center, Wroclaw, Lower Silesian Voivodeship, Poland
- Spain (2):
  - Public Health Directorate, SERGAS, Santiago de Compostela, Galicia
  - Althaia Foundation, Manresa

IPD SHARING:
Plan to Share IPD: No
Individual Patient Data data sharing is not foreseen in the informed consent form, however, de-identified patient data will be shared for research purposes.

REFERENCES:
- See also: Links to all PRAISE U publications — https://uroweb.org/praise-u/news